CLINICAL TRIAL: NCT05566093
Title: Endoscopic Ultrasound-guided Fine-needle Injection for Nonfunctional Pancreatic Neuroendocrine Tumors: a Prospective Multicenter Study
Brief Title: EUS-FNI for Nonfunctional Pancreatic Neuroendocrine Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Shanyu Qin, Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K039-01
Record Dates: First submitted 2022-09-25; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Nonfunctional Pancreatic Neuroendocrine Tumor; Pancreatic Neuroendocrine Tumor; Endoscopic Ultrasound
Keywords: Nonfunctional Pancreatic Neuroendocrine Tumor; Endoscopic ultrasonography-guided fine-needle injection; Ablation; Endoscopic ultrasonography
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor; Adenoma, Islet Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nonfunctional pancreatic neuroendocrine tumors (Experimental): The patients with NF-pNETs will undergo EUS-guided ethanol or lauromacrogol ablation
  Interventions: Procedure: EUS-guided ethanol ablation; Procedure: EUS-guided lauromacrogol ablation

INTERVENTIONS:
Procedure: EUS-guided ethanol ablation — After puncturing with the needle, 95% ethanol under the guidance of EUS was injected into the tumor. The injection volume of ethanol was estimated according to the following principles: (1) The injection volume was not larger than the tumor spherical volume. (2) Injection volume was reduced when the tumor was adjacent to the pancreatic duct or vessel. (3) Injection volume for the lesions with repeated EUS-FNI was reduced.
Procedure: EUS-guided lauromacrogol ablation — After puncturing with the needle, lauromacrogol under the guidance of EUS was injected into the tumor. The injection volume of lauromacrogol was estimated according to the following principles: (1) The injection volume was not larger than the tumor spherical volume. (2) Injection volume was reduced when the tumor was adjacent to the pancreatic duct or vessel. (3) Injection volume for the lesions with repeated EUS-FNI was reduced.

SUMMARY:
The current study aims to access the feasibility, safety, and efficacy of EUS-FNI for nonfunctional pNETs

DETAILED DESCRIPTION:
The management of nonfunctional pancreatic neuroendocrine tumors (NF-pNETs) remains controversial. In general, surgical resection is the standard treatment for NF-pNETs. However, the incidence of postoperative adverse events of surgical resection is relatively high. Recently, several studies have revealed that endoscopic ultrasonography (EUS)-guided fine-needle injection (EUS-FNI) with ethanol or lauromacrogol may offer an effective treatment for pNETs. Therefore, a multicenter prospective study is being conducted to further identify the efficacy and safety of EUS-FNI for NF-pNETs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with NF-pNETs are evaluated by cytology or immunohistochemistry.
2. Patients who refuse surgery or observation.
3. Patients who have given their fully informed consent.

Exclusion Criteria:

1. Patients who are not suitable for EUS-FNI.
2. Patients who have poor conditions including blood coagulation dysfunction, mental disorders, and mild or severe cardiorespiratory.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of complete ablation | At 24 months after treatment
  The rate of complete ablation on the CE-CT or CE-EUS
The Chang The change of tumor size | From baseline to 24 months
  The change of tumor size on the CE-CT or EUS

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Within 3 month after treatment
  The incidence of adverse events （such as abdominal pain, hematoma formation, ulcer at the puncture site, acute pancreatitis, pancreatic necrosis, and pancreatic duct stricture）

CONTACTS AND LOCATIONS:
Overall Officials: Shanyu Qin, MD,Ph.D, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes